CLINICAL TRIAL: NCT04019626
Title: An Open-label, Parallel Study to Assess Tobacco-related Biomarkers of Exposure, Biomarkers of Potential Harm, and Nicotine Uptake During a 56-day Switch to Myblu E-cigarettes in Adult Smokers
Brief Title: A Study to Assess Tobacco-related Biomarkers of Exposure in Smokers Using myBlu E-cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fontem Ventures BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CA22747
Record Dates: First submitted 2019-07-12; First posted 2019-07-15 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Continue-smoking (Active Comparator): The subject's usual brand of combustible cigarette
  Interventions: Other: Continue-smoking
- myblu Tobacco 2.5% (Experimental): myblu e-cigarette system with Tobacco flavor, 2.5% nicotine. At Day 28 of the study, subjects may be allowed to switch to another myblu variant.
  Interventions: Other: myblu Tobacco 2.5%
- myblu Tobacco 4.0% (Experimental): myblu e-cigarette system with Tobacco flavor, 4.0% nicotine. At Day 28 of the study, subjects may be allowed to switch to another myblu variant.
  Interventions: Other: myblu Tobacco 4.0%
- myblu Honeymoon 2.5% (Experimental): myblu e-cigarette system with Honeymoon flavor, 2.5% nicotine. At Day 28 of the study, subjects may be allowed to switch to another myblu variant.
  Interventions: Other: myblu Honeymoon 2.5%
- myblu Honeymoon 4.0% (Experimental): myblu e-cigarette system with Honeymoon flavor, 4.0% nicotine. At Day 28 of the study, subjects may be allowed to switch to another myblu variant.
  Interventions: Other: myblu Honeymoon 4.0%
- JUUL 5% (Active Comparator): JUUL® system with Virginia Tobacco Flavor JUULpod, 5.0% nicotine. This arm is only included in the PK sub-study.
  Interventions: Other: JUUL 5%

INTERVENTIONS:
Other: Continue-smoking — Ad-libitum use of subjects' usual brand combustible cigarette
  Arms: Continue-smoking
Other: myblu Tobacco 2.5% — Ad-libitum use of myblu e-cigarette with Tobacco flavor 2.5% nicotine
  Arms: myblu Tobacco 2.5%
Other: myblu Tobacco 4.0% — Ad-libitum use of myblu e-cigarette with Tobacco flavor 4.0% nicotine
  Arms: myblu Tobacco 4.0%
Other: myblu Honeymoon 2.5% — Ad-libitum use of myblu e-cigarette with Honeymoon flavor 2.5% nicotine
  Arms: myblu Honeymoon 2.5%
Other: myblu Honeymoon 4.0% — Ad-libitum use of myblu e-cigarette with Honeymoon flavor 4.0% nicotine
  Arms: myblu Honeymoon 4.0%
Other: JUUL 5% — Ad-libitum use of JUUL 5% e-cigarette
  Arms: JUUL 5%

SUMMARY:
The purpose of this study is to assess changes in exposure to selected harmful and potentially harmful substances related to tobacco/nicotine use when adult smokers switch from their usual brand of combustible cigarettes to the myblu e-cigarette, for up to 56 days. This study is designed as an open-label, partially-randomized, parallel-arm, multi-site study in healthy adult smokers.

Some subjects will be selected to take part in additional procedures as part of a pharmacokinetics (PK) sub-study.

DETAILED DESCRIPTION:
Subjects are randomized to either continue smoking conventional cigarettes, or switch to use the myblu e-cigarette. Within the "myblu" arm, subjects were assigned to one of four variants of the myblu e-cigarette, having different flavors and nicotine strengths. Initial product assignment for each subject was based on preference as a method to enhance compliance. To further improve compliance through Day 56, subjects may have been allowed to choose to switch to another variant of the myblu e-cigarette, or to continue using the same e-liquid selected initially.

ELIGIBILITY:
Inclusion Criteria:

* Having smoked ≥5 manufactured combustible cigarettes per day for at least one year
* Exhaled carbon monoxide level of >10 ppm at screening
* Tested positive for urinary cotinine (approximately 200 ng/mL) at screening

Exclusion Criteria:

* Relevant illness history
* Relevant medication use
* Body mass index (BMI) of less than 18 kg/m2 or greater than 40 kg/m2
* Allergy to propylene glycol or glycerin
* Use of nicotine-containing products other than manufactured cigarettes
* Use of prescription smoking cessation treatments
* Smokers who draw smoke into their mouth and throat but do not inhale
* Intent or desire to stop smoking
* Female subjects who are pregnant, lactating, or intend to become pregnant

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Myblu Tobacco Flavor 2.5%: Use of myblu e-cigarette system with tobacco flavor 2.5% nicotine
- Myblu Tobacco Flavor 4.0%: Use of myblu e-cigarette system with tobacco flavor 4.0% nicotine
- Myblu Honeymoon 2.5%: Use of myblu e-cigarette system with Honeymoon flavor 2.5% nicotine
- Myblu Honeymoon 4.0%: Use of myblu e-cigarette system with Honeymoon flavor 4.0% nicotine
- JUUL 5%: Use of JUUL 5% nicotine e-cigarette
Period: Overall Study
Arm/Group | Myblu Tobacco Flavor 2.5% | Myblu Tobacco Flavor 4.0% | Myblu Honeymoon 2.5% | Myblu Honeymoon 4.0% | Continue-smoking | JUUL 5%
Started | 42 | 42 | 45 | 46 | 44 | 21
Completed | 36 | 32 | 37 | 39 | 38 | 20
Not Completed | 6 | 10 | 8 | 7 | 6 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: randomized subjects in the main study with at least one documented product-use experience from Day 1. The JUUL5% arm is not included as it was used only for the PK sub-study as a secondary objective, and not the main study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Myblu Tobacco Flavor 2.5% | Myblu Tobacco Flavor 4.0% | Myblu Honeymoon 2.5% | Myblu Honeymoon 4.0% | Continue-smoking | Total
Number analyzed (Participants) | 42 | 42 | 45 | 46 | 44 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (11.72) | 37.8 (10.47) | 40.3 (9.43) | 40.3 (9.75) | 39.7 (10.44) | 39.6 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 18 | 20 | 18 | 84
  Male | 28 | 28 | 27 | 26 | 26 | 135
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 12 | 16 | 18 | 16 | 13 | 75
  White | 27 | 23 | 24 | 27 | 30 | 131
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 3 | 1 | 1 | 9
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (4.7) | 30.0 (4.9) | 28.9 (4.7) | 28.9 (5.2) | 29.9 (5.6) | 29.1 (5.1)
Blood carboxyhemoglobin (COHb) % [Mean (Standard Deviation); unit: % saturation] | 4.9 (2.2) | 4.8 (1.8) | 4.8 (2.1) | 5.3 (1.9) | 5.7 (2.0) | 5.1 (2.0)
4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) amount excreted in urine [Mean (Standard Deviation); unit: ng/24 hours] — Population: Some samples were missing
  ng/24 hours
    number analyzed (Participants) | 42 | 42 | 41 | 45 | 44 | 214
    (all) | 411.0 (333.2) | 406.8 (328.8) | 410.4 (351.2) | 479.4 (404.2) | 513.7 (403.7) | 444.26 (346.2)
3-hydroxypropylmercapturic acid (3-HPMA) amount excreted in urine [Mean (Standard Deviation); unit: ug/24 hours] — Population: Some samples were missing
  ug/24 hours
    number analyzed (Participants) | 42 | 42 | 41 | 45 | 44 | 214
    (all) | 1592.5 (818.2) | 1730.3 (1044.2) | 1749.7 (780.1) | 1919.0 (999.8) | 2214.0 (1172.6) | 1841.1 (963.0)
S-phenyl mercapturic acid (S-PMA) amount excreted in urine [Mean (Standard Deviation); unit: ug/24 hours] — Population: Some samples were missing
  ug/24 hours
    number analyzed (Participants) | 42 | 42 | 41 | 45 | 44 | 214
    (all) | 5.3 (3.7) | 5.9 (4.3) | 6.5 (5.1) | 7.2 (5.2) | 8.6 (5.9) | 6.7 (4.8)
Nicotine equivalents amount excreted in urine [Mean (Standard Deviation); unit: mg/24 hours] — Population: Some samples were missing
  mg/24 hours
    number analyzed (Participants) | 42 | 42 | 41 | 45 | 44 | 214
    (all) | 13.6 (6.8) | 14.1 (7.5) | 17.1 (13.3) | 16.2 (6.5) | 18.0 (7.3) | 15.8 (8.3)
Level of white blood cells [Mean (Standard Deviation); unit: cells*thousands/uL] — Population: Some samples were missing
  cells*thousands/uL
    number analyzed (Participants) | 42 | 40 | 45 | 46 | 44 | 217
    (all) | 7.7 (2.0) | 7.0 (2.0) | 6.8 (1.8) | 7.4 (2.0) | 7.2 (2.2) | 7.2 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Carboxyhemoglobin in Blood
Description: Change from baseline in the % saturation of carboxyhemoglobin (COHb) in whole blood
Time Frame: Baseline and 56 days
Population: Available data from the Intent-to-treat population (ITT; randomized subjects in the main study with at least one documented product-use experience from Day 1) is presented. Subjects using the myblu e-cigarette were allowed to switch product variant in the course of the study (cf "Study Description"). Therefore, the number of subjects analysed in one arm may be different from the number of subjects who were initially assigned to this product at the study start. JUUL arm was only for PK sub-study
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Myblu Tobacco Flavor 2.5% | Myblu Tobacco Flavor 4.0% | Myblu Honeymoon 2.5% | Myblu Honeymoon 4.0% | Continue-smoking
Number analyzed (Participants) | 32 | 49 | 24 | 33 | 37
% change from baseline | -59.6 (23.3) | -62.7 (19.4) | -46.4 (35.1) | -62.7 (21.2) | 8.5 (28.3)

2. Primary Outcome: Amount of 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol in Urine in 24 Hours
Description: Change from baseline in the amount of 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL - a biomarker of exposure to 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone) excreted in urine in 24-hours
Time Frame: Baseline and 56 days
Population: Available data from the Intent-to-treat population (ITT; randomized subjects in the main study with at least one documented product-use experience from Day 1) is presented. Subjects using the myblu e-cigarette were allowed to switch product variant in the course of the study (see "Study Description"). Therefore, the number of subjects analysed in one arm may be different than the number of subjects who were initially assigned to this product at the study start. JUUL arm was only for PK sub-study
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Myblu Tobacco Flavor 2.5% | Myblu Tobacco Flavor 4.0% | Myblu Honeymoon 2.5% | Myblu Honeymoon 4.0% | Continue-smoking
Number analyzed (Participants) | 32 | 52 | 25 | 35 | 38
% change from baseline | -58.3 (72.8) | -44.7 (150.5) | -62.7 (36.2) | -70.7 (33.7) | 1.1 (29.6)

3. Primary Outcome: Amount of 3-hydroxypropylmercapturic Acid in Urine in 24 Hours
Description: Change from baseline in the amount of 3-hydroxypropylmercapturic acid (3-HPMA - a biomarker of exposure to acrolein) excreted in urine in 24-hours
Time Frame: Baseline and 56 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Myblu Tobacco Flavor 2.5% | Myblu Tobacco Flavor 4.0% | Myblu Honeymoon 2.5% | Myblu Honeymoon 4.0% | Continue-smoking
Number analyzed (Participants) | 32 | 52 | 25 | 35 | 38
% change from baseline | -60.0 (28.2) | -55.7 (46.1) | -50.5 (36.2) | -53.8 (64.5) | 1.6 (40.6)

4. Primary Outcome: Amount of S-phenyl Mercapturic Acid in Urine in 24 Hours
Description: Change from baseline in the amount of s-phenyl mercapturic acid (S-PMA - a biomarker of exposure to benzene) excreted in urine in 24-hours
Time Frame: Baseline and 56 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Myblu Tobacco Flavor 2.5% | Myblu Tobacco Flavor 4.0% | Myblu Honeymoon 2.5% | Myblu Honeymoon 4.0% | Continue-smoking
Number analyzed (Participants) | 32 | 52 | 25 | 35 | 38
% change from baseline | -85.9 (32.5) | -44.9 (257.5) | -63.1 (79.3) | -73.8 (55.7) | -2.7 (38.4)

5. Secondary Outcome: Amount of Nicotine Equivalents in Urine in 24 Hours
Description: The change from baseline in the amount of nicotine equivalents excreted in urine in 24-hours
Time Frame: Baseline and 56 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Myblu Tobacco Flavor 2.5% | Myblu Tobacco Flavor 4.0% | Myblu Honeymoon 2.5% | Myblu Honeymoon 4.0% | Continue-smoking
Number analyzed (Participants) | 32 | 51 | 24 | 35 | 38
% change from baseline | -7.8 (74.0) | 16.6 (61.1) | -13.8 (54.5) | -1.3 (38.8) | -7.0 (27.0)

6. Secondary Outcome: Level of White Blood Cells
Description: The change from baseline in the level of white blood cells, which is a biomarker of potential harm
Time Frame: Baseline and 56 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Myblu Tobacco Flavor 2.5% | Myblu Tobacco Flavor 4.0% | Myblu Honeymoon 2.5% | Myblu Honeymoon 4.0% | Continue-smoking
Number analyzed (Participants) | 31 | 51 | 25 | 35 | 37
% change from baseline | -9.2 (16.7) | -4.3 (16.8) | -8.7 (17.9) | -8.5 (16.3) | 4.7 (17.0)

7. Secondary Outcome: Subjective Measure: Nicotine Withdrawal Symptoms Total Score
Description: Nicotine withdrawal symptoms are measured using the Minnesota Tobacco Withdrawal Scale-Revised (MTWS-R) questionnaire. The DSM-5 and craving items from the MTWS-R have been included. The subjects rate themselves on the questionnaire, which includes symptoms such as angry, irritable, frustrated, depressed mood, restless, insomnia. Each question is rated from 0 (none) to 4 (severe). Total scores may range from 0 to a maximum of 32.
Time Frame: 56 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Myblu Tobacco Flavor 2.5% | Myblu Tobacco Flavor 4.0% | Myblu Honeymoon 2.5% | Myblu Honeymoon 4.0% | Continue-smoking
Number analyzed (Participants) | 31 | 51 | 26 | 33 | 38
score on a scale | 8.6 (6.7) | 5.7 (5.5) | 7.1 (5.3) | 6.8 (5.8) | 8.1 (5.9)

8. Secondary Outcome: Maximum Nicotine Concentration in Blood
Description: The maximum nicotine concentration in blood (Cmax)
Time Frame: 5 minutes prior, and at 3, 5, 7, 10, 12, 15, 20, 30, 60, 120 and 180 minutes post dose
Population: Sub-group of participants who participated in the PK sub-study, on Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- JUUL® 5.0%: Use of JUUL® system with Virginia Tobacco Flavor JUULPod, 5.0% nicotine
Arm/Group | Myblu Tobacco Flavor 2.5% | Myblu Tobacco Flavor 4.0% | Myblu Honeymoon 2.5% | Myblu Honeymoon 4.0% | Continue-smoking | JUUL® 5.0%
Number analyzed (Participants) | 20 | 19 | 19 | 22 | 24 | 19
ng/mL | 4.0 (196.3) | 7.3 (118.6) | 4.3 (191.3) | 8.9 (159.8) | 13.5 (62.5) | 6.9 (160.1)

ADVERSE EVENTS:
Time Frame: 72 days (58 study days plus 14 follow-up days) for all arms except JUUL. 15 day for JUUL arm.
Description: Adverse events of the Safety Population (all subjects with at least one reported product use from Day -1) is presented. Subjects using the myblu e-cigarette were allowed to switch product variant in the course of the study (see "Study Description"). Therefore, the number of subjects at risk in one arm may be different than the number of subjects who were initially assigned to this product at the study start.
Arm/Group | Myblu Tobacco Flavor 2.5% | Myblu Tobacco Flavor 4.0% | Myblu Honeymoon 2.5% | Myblu Honeymoon 4.0% | Continue-smoking | JUUL® 5.0%
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/71 | 0/47 | 0/57 | 0/44 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/71 | 0/47 | 0/57 | 0/44 | 0/21
Other Adverse Events (participants affected / at risk) | 8/55 | 10/71 | 6/47 | 6/57 | 7/44 | 8/21
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myblu Tobacco Flavor 2.5% (N=55) | Myblu Tobacco Flavor 4.0% (N=71) | Myblu Honeymoon 2.5% (N=47) | Myblu Honeymoon 4.0% (N=57) | Continue-smoking (N=44) | JUUL® 5.0% (N=21)
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 2 | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 4 | 2 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT04019626/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT04019626/SAP_001.pdf